CLINICAL TRIAL: NCT01517217
Title: Randomised Trial Evaluating the Effect of Postoperative Girdle Following Major Abdominal Surgery
Brief Title: Effect of Postoperative Girdle Following Abdominal Surgery on Pulmonary Function, Mobilisation and Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Karin Strigard, ass. professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20110201KI
Record Dates: First submitted 2012-01-09; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Pain, Postoperative; Respiratory Depression
Keywords: girdle; laparotomy; pulmonary function; postoperative pain; mobilisation
MeSH Terms: conditions — Pain, Postoperative; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No girdle postoperative (Other): patients undergoing major abdominal surgery will get NO individualized girdle. Functional outcomes as pulmonary function and pain are measured daily. Participants will be followed for the duration of 5 days or the duration of hospital stay, if shorter than 5 days.
  Interventions: Procedure: No girdle
- Girdle postoperative (Other): patients undergoing major abdominal surgery will get an individualized girdle. Functional outcomes as pulmonary function and pain are measured daily. Participants will be followed for the duration of 5 days or the duration of hospital stay, if shorter than 5 days.
  Interventions: Procedure: Girdle

INTERVENTIONS:
Procedure: No girdle — No girdle is used for the first five postoperative days
  Arms: No girdle postoperative
Procedure: Girdle — Girdle the first five postoperative days
  Arms: Girdle postoperative

SUMMARY:
There is a considerable lack of knowledge in everyday surgical practice concerning treatment with a corset after laparotomy, in surgery for incisional hernia or as conservative treatment.

The aims are to elucidate effects of corset treatment on patient experience and pain, physiology and abdominal wall strength.

Effects of corset treatment after laparotomy will be studied in a randomised trial with the hypothesis that postoperative corset-use improves respiratory physiology and reduce pain. The primary end-point is PeakCoughFlow change, secondary end-points are vital capacity, residual volumes and patient perception as measured by the ventral hernia pain questionnaire (VHPQ) developed by our group. This study is powered for 50 patients.

Conclusions from the study are of such a nature that they can be immediately transferred to clinical practice.

DETAILED DESCRIPTION:
Presently, there is a significant lack of knowledge in everyday surgical practice concerning treatment for incisional hernias and treatment with a corset before and after surgery or as a means of conservative treatment. For many years, corsets have been used in surgical departments without evidence to support this practice.

Corsets are expensive and require good patient compliance. Some arguments for the use of corsets are reduced pain and tension in the abdominal wall and prevention of the development and recurrence of incisional hernias, as well as their use as a truss in cases where conservative treatment is decided on.

The aim of this project is thus to ameliorate the lack of knowledge surrounding corset use.

More specifically, the aims of the project are to clarify the effects of corset use on

1. Physiological parameters

   * Measured with spirometry, Vital capacity (VC), Forced Expiratory Volume (FEV), Peak Expiratory Flow (PEF) and with coughPEF
2. Patient comfort, pain and self-perceived experience

   * Measured with VAS scale for pain. VHPQ (ventral hernia pain questionary) for pain. Recording of medication. Grade of mobilisation.

Corset treatment has been thought to affect cardiovascular and respiratory function as well as intra abdominal pressure both in positive and negative directions. There are no scientific publications that specifically describe and evaluate these effects. One reason for this could be that the assessment of such parameters is difficult and time-consuming in clinical practice, for instance spirometry. Less complicated alternatives e.g. Peak Expiratory Flow rate (PEF) has been considered too imprecise. However, recently, a simpler and more efficient instrument has been developed for measuring lung function, the Peak Cough Flow (PCF). It has been validated for use in pulmonary function testing in patients with neuromuscular disorders, where it is used to predict the risk of an inadequate coughing response and mucus clearance. Moreover, portable digital spirometers have been developed that can be easily used in an ambulatory setting. Postoperatively, similar problems may arise with a reduction in vital capacity. It is therefore important to investigate the effects of corsets on lung function.

Many patients that undergo laparotomy have an indwelling urinary catheter during the first postoperative days, often as a result of epidural anaesthesia but also for monitoring of fluid balance. A urinary catheter also allows for the measurement of the intra abdominal pressure, which, together with the measurement of systemic blood pressure, gives a good estimate of physiological parameters which can be used to compare different treatment groups.

A randomised controlled study concerning the postoperative use of corsets after laparotomy.

Hypothesis: Postoperative corset-use improves respiratory physiology as measured using the PCF without impairing other spirometric parameters. Corsets also reduce pain and discomfort after surgery.

Consecutive patients undergoing laparotomy at the Centre for Gastrointestinal surgery at the Karolinska University Hospital are asked whether they would accept to participate in a randomised study where one arm receives a corset for five days postoperatively and the other does not receive a corset after laparotomy. The primary end-point is PCF change, secondary end-points are vital capacity, residual volumes and patient perception as measured by the VHPQ. A GCP-trained research nurse with extensive experience will be in charge of monitoring and collection of data. PCF will be measured using a portable PCF apparatus (Peak flow meter, HS Clerment Clarke International) whereas other spirometric parameters are measured using a portable computer-assisted vitalograph (IM-Medico ML 2525). Pain and the functional status of the patients will be measured using the VHPQ as described above and the EuroQoL.

Based on previous measurements, a normal PCF without corset is assumed to be around 360ml/min. Assuming that the standard deviation is 40ml/min and that the corset improves performance by 10%, 21 patients will be required in each group (42 in total) at 95% significance level and power of 80%. In order to compensate for patient drop-out, we plan to include 50 patients. If intra abdominal pressure rises above 28cmH2O or if there are signs of wound infection, the corset will be removed. The wound will be photographed on day five in all patients.

ELIGIBILITY:
The inclusion in the study is done to reflect the normal population on a colorectal surgery ward.

Inclusion Criteria:

* Patients undergoing laparotomy with a midline incision more than 12 cm
* Over 18 years of age
* Planned time at ward less than 10 days
* Not on oxygen treatment at home

The exclusion criteria are minimized but made to avoid obvious confounding

Exclusion Criteria:

* Dementia
* Not possible to understand instructions
* Children (<18 years of age)
* Not involved in other studies during the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
pulmonary function | 20120630
  Participans will be followed for the duration of 5 days or the duration of hospital stay, if shorter than 5 days. Spirometry will be assessed the day before surgery and therafter the day after surgery and every day after the end of the study.

SECONDARY OUTCOMES:
postoperative pain | 20120630
  pain meassured with VAS scale and amount of medication

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, ass prof, Principal Investigator — Karolinska Institutet; Leonard Clay, Dr, Study Chair — Karolinska Institutet; Ulf Gunnarsson, Prof, Study Director — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Clay L, Gunnarsson U, Franklin KA, Strigard K. Effect of an elastic girdle on lung function, intra-abdominal pressure, and pain after midline laparotomy: a randomized controlled trial. Int J Colorectal Dis. 2014 Jun;29(6):715-21. doi: 10.1007/s00384-014-1834-x. Epub 2014 Jan 28. PMID 24468797